CLINICAL TRIAL: NCT00799825
Title: Safety Study of GSK Biologicals' Human Papillomavirus Vaccine (GSK580299) in Female American and Canadian Subjects Who Had Received Control Vaccine in Study 580299/008
Brief Title: Safety Study of GSK Biologicals' Human Papillomavirus Vaccine in 580299/008 Subjects From Canada or the US
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111955
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2013-09-20 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Infections, Papillomavirus
Keywords: papillomavirus; HPV vaccine; cervical cancer; HPV; human papillomavirus
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (1):
- Cervarix group (Experimental): Female subjects who previously received the active control i.e. Hepatitis A vaccine in the primary study (NCT00122681) and who received the Cervarix vaccine in the current study. The Cervarix vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm according to a 0, 1 and 6 months schedule.
  Interventions: Biological: GSK Biological's HPV vaccine GSK580299 (Cervarix™)

INTERVENTIONS:
Biological: GSK Biological's HPV vaccine GSK580299 (Cervarix™) — All subjects will receive a 0.5 ml dose administered as an intramuscular injection, according to a 0, 1, 6-month schedule.
  Other Names: CervarixTM

SUMMARY:
This phase 3b study is designed to assess the safety of GlaxoSmithKline Biological's HPV vaccine GSK580299 in female subjects who took part in study 580299/008 and received the control vaccine (Hepatitis A vaccine).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study
* A subject previously enrolled in the primary study (NCT00122681), who received the active control hepatitis A vaccine, and who cannot receive commercially available HPV-16/18 L1 VLP AS04 vaccine because the vaccine has not yet been granted licensure in the subject's country or because the subject is above the age for which the vaccine is licensed.
* Written informed consent must be obtained from the subject prior to enrolment.
* A woman aged 18 years or older, at the time of the first vaccination in this study.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must not be pregnant. Absence of pregnancy should be verified with a urine pregnancy test.
* Subject must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Pregnant or lactating female. Enrolment should be deferred until three months after pregnancy has been completed or after lactating has ceased.
* A woman planning to become pregnant or likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive prevention during the study period and up to two months after the last vaccine dose.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and the extended safety follow-up period.
* Concurrently participating in another clinical study at any time during the study period, in which the subject has been or will be exposed to an investigational or non-investigational product (pharmaceutical product or device).
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study other than that foreseen by protocol.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days (i.e. Day 0-29) of each dose of vaccine. Administration of routine meningococcal, hepatitis B, hepatitis A, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before each dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Previous administration of components of the investigational vaccine.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccine.
* Hypersensitivity to latex.
* Acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, haematological, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests, which in the opinion of the investigator precludes administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Cancer or autoimmune disease under treatment.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Acute disease at the time of enrolment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2009-01-01; Primary Completion 2012-08-02 (Actual); Study Completion 2012-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (37):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Louisville, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, New Bern, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pleasant Hills, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Canada (9):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Beauport, Quebec
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects in this study come from the primary study (NCT00122681) where they were included in the control group and received Hepatitis A vaccination. The number of subjects that started the study included only those subjects with the vaccine dose administered.
Period: Overall Study
Arm/Group | Cervarix Group
Started | 344
Completed | 296
Not Completed | 48
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 38
Not completed — Pregnancy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 344
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.4 (2.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 344
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Any = Occurrence of any SAE regardless of intensity grade or relation to vaccination. Grade 3 = SAE which prevented normal, everyday activities. Related = SAE assessed by the investigator as related to the vaccination.
Time Frame: Throughout the study (up to Month 12)
Population: The analyses were performed on the Total Vaccinated cohort, which included all subjects who received at least one dose of Cervarix vaccine in this study, for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 344
Subjects
  Any SAEs | 8
  Grade 3 SAEs | 5
  Related SAEs | 0

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Medically Significant Conditions (MSCs)
Description: MSCs = Adverse events (AEs) prompting emergency room/physician visits not related to common diseases or routine visits for physical examination/vaccination, or SAEs not related to common diseases. Common diseases include: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury. Any = Occurrence of any MSC regardless of intensity grade or relation to vaccination. Grade 3 = MSC which prevented normal, everyday activities. Related = MSC assessed by the investigator as related to the vaccination.
Time Frame: Throughout the study (up to Month 12)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 344
Subjects
  Any MSCs | 32
  Grade 3 MSCs | 9
  Related MSCs | 0

3. Primary Outcome: Number of Subjects With Pregnancies and Pregnancy Outcomes.
Time Frame: Throughout the study (up to Month 12)
Population: The analysis was based on pregnant subjects from the Total Vaccinated cohort, which included all subjects who received at least one dose of Cervarix vaccine in this study, for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 19
Subjects
  Live infant NO apparent congenital anomaly | 14
  Elective termination NO apparent congenital anom. | 2
  Spontaneous abortion NO apparent congenital anom. | 2
  Lost to follow up | 1

ADVERSE EVENTS:
Time Frame: SAEs were reported throughout the study period, from Day 0 up to Month 12.
Description: No other adverse events were reported.
Arm/Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 8/344
Other Adverse Events (participants affected / at risk) | 0/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=344)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.